CLINICAL TRIAL: NCT01202175
Title: Effects of the Novel Beta-adrenergic Antagonist Nebivolol (Bystolic) on Prehypertensive Subjects at Genetic Risk of Hypertension: Implications for Inflammation, Endothelial Dysfunction, and Oxidative Stress.
Brief Title: Effects of the Beta-blocker Nebivolol (Bystolic) on Subjects With High Normal Blood Pressure and/or a Family History of Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Joachim H. Ix, Professor of medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100353
Record Dates: First submitted 2010-06-24; First posted 2010-09-15 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-07

CONDITIONS: Pre-hypertension; Hypertension
Keywords: Genetic risk of hypertension
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Nebivolol (Experimental)
  Interventions: Drug: Nebivolol
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Oral nebivolol 2.5-5mg once daily
  Other Names: Bystolic

SUMMARY:
The investigators aim to evaluate subjects at high risk of future development of hypertension, those with a family history of hypertension and/or that already have high normal(SBP 120-139 mmHg or DBP 80-89 mmHg) blood pressure. The investigators plan to investigate whether these subjects have the same markers (such as microscopic protein in the urine or C-reactive protein in the blood) in the blood and urine that people with high blood pressure have, and whether they are improved before and after taking the beta-blocker nebivolol.

ELIGIBILITY:
Inclusion Criteria:

* • Prehypertensive male and female subjects with SBP =120-139 or DBP =80-89 with at least one known family member (must be diagnosed prior to the age of 60) with essential hypertension (confirmation may be sought).

  * All ethnicities
  * Non-smokers and non-drug abusers, no current smoking or illicit drug use in the prior 3 months.
  * Aged 18-40 years
  * No known serious medical conditions requiring close monitoring from physicians- such as liver impairment, chronic kidney disease, or diabetes mellitus
  * Subjects will need to remain in the San Diego area for the duration of the study (10 weeks) and be accessible by telephone or email.
  * Female subjects must be willing to use a birth control method, such as abstinence, birth control pills, diaphragm, condom, or intrauterine device to prevent pregnancy during the study.

Exclusion Criteria:

* Subjects with SBP >140 or SBP<120 or DBP >90 and DBP<80
* We will exclude subjects whose family members have known secondary etiologies for hypertension such as hyperaldosteronism or Cushing's Disease.
* Subjects cannot have a chronic medical condition that is actively treated by a physician, such as liver impairment, diabetes, or kidney disease
* History of bronchial asthma or chronic obstructive pulmonary disease
* Subjects cannot be on any anti-hypertensive medications for any reason.
* Subjects may not have previous intolerance, hypersensitivity, or allergy to any beta blocker therapy or may have contraindications to beta blocker therapy such as asthma, bradycardia, etc.
* Subjects may not be taking medications which may affect the metabolism of nebivolol, such as those that inhibit CYP2D6 (such as fluoxetine or cimetidine)
* Nursing women, pregnant women, or those that plan to become pregnant in the study period will also be excluded. (Pregnancy tests will be performed on all female subjects at the start of the study)
* Subjects with pulse rate consistently <60 beats per minute or evidence of arrythmias including atrioventricular block.
* Those that have smoked or used illicit drugs within the past 3 months
* Female subjects that are not willing to use a birth control method, such as abstinence, birth control pills, diaphragm, condom, or intrauterine device to prevent pregnancy during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O'Connor, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study results are being entered according to a publication that was published before PI passed away. According to the publication; two participants dropped out because of flu-like symptoms, 2 were lost to follow-up, and 1 dropped out of the study after the initial visit but never took the medication. It is unknown what arm they were in.
Groups:
- All Study Participants: Oral nebivolol 5 mg once daily or Placebo (sugar pill) once dailly. Arms/Groups are combined in this module because the only access to data is a publication that was published before Principal Invesitgator passed away. According to the publication; two participants dropped out because of flu-like symptoms, 2 were lost to follow-up, and 1 dropped out of the study after the initial visit but never took the medication. It is unknown what arm they were in.
Period: Overall Study
Arm/Group | All Study Participants
Started | 50
Nebivolol | 25
Pacebo | 25
Completed | 45
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Nebivolol: Nebivolol: Oral nebivolol 5 mg once daily
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (1.8) | 30.4 (1.6) | 33.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 18 | 12 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 3 | 9
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.55 (0.92) | 31.03 (1.14) | 29.79 (.86)
Starting systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 127.4 (1.6) | 126.2 (1.5) | 126.8 (1.1)
Starting diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 84.7 (1.5) | 84.4 (1.0) | 84.5 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Aortic Systolic Blood Pressure (SBP)
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
mm Hg
  Baseline (visit 1) | 112.7 (2.5) | 107.7 (1.9)
  Week 8 (visit 2) | 106.2 (2.4) | 106.6 (2.0)

2. Primary Outcome: Aortic Diastolic Blood Pressure (DBP)
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
mm Hg
  Baseline (visit 1) | 79.1 (2.3) | 75.9 (1.7)
  Week 8 (visit 2) | 71.3 (1.9) | 74 (1.8)

3. Primary Outcome: Aortic Mean Arterial Pressure (MAP)
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
mm Hg
  Baseline (visit 1) | 94.2 (2.1) | 90.4 (1.6)
  Week 8 (visit 2) | 86.8 (1.9) | 88.6 (1.9)

4. Primary Outcome: Aortic Pulse Pressure
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
mm Hg
  Baseline (visit 1) | 33.6 (2.3) | 31.8 (1.4)
  Week 8 (visit 2) | 34.9 (1.8) | 32.6 (1.2)

5. Primary Outcome: Aortic Augmentation Pressure
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
mm Hg
  Baseline (visit 1) | 7.4 (2.0) | 5.5 (1.0)
  Week 8 (visit 2) | 6.8 (1.6) | 5.3 (1.1)

6. Primary Outcome: Aortic Augmentation Index for Heart Rate
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
percentage
  Baseline (visit 1) | 14.7 (3.4) | 14.5 (2.4)
  Week 8 (visit 2) | 11.9 (3.8) | 12.8 (2.9)

7. Primary Outcome: Pulse Wave Velocity
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
m/s
  Baseline (visit 1) | 6.73 (0.28) | 5.95 (0.19)
  Week 8 (visit 2) | 6.00 (0.18) | 5.78 (0.19)

8. Primary Outcome: Heart Rate, Beats Per a Minute
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: beats per a minute
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
beats per a minute
  Baseline (visit 1) | 72.0 (1.9) | 75.6 (1.9)
  Week 8 (visit 2) | 64.4 (2.3) | 72.1 (2.0)

9. Secondary Outcome: Urinary Nitric Oxide Excretion
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: umol/ mg Cr
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
umol/ mg Cr
  Baseline (visit 1) | 40.31 (5.05) | 61.77 (11.86)
  Week 8 (visit 2) | 64.38 (14.25) | 65.54 (10.54)

10. Secondary Outcome: Urinary Isoprostane Excretion
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: pg/ mg Cr
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
pg/ mg Cr
  Baseline (visit 1) | 180 (14) | 165 (17)
  Week 8 (visit 2) | 213 (20) | 185 (22)

11. Secondary Outcome: Urinary Hydrogen Peroxide Excretion
Time Frame: Baseline (visit 1) and 8 Weeks (visit 2)
Measure: Mean (Standard Error); unit: umol/ mg Cr
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
umol/ mg Cr
  Baseline (visit 1) | 0.652 (0.274) | 0.500 (0.281)
  Week 8 (visit 2) | 2.79 (1.83) | 0.578 (0.194)

12. Secondary Outcome: Plasma Interleukin Levels
Time Frame: Basline (visit 1) and 8 weeks (visit 2)
Measure: Mean (Standard Deviation); unit: pg/ mL
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 25 | 25
pg/ mL
  Baseline (visit 1) | 1.626 (0.598) | 1.351 (0.258)
  Week 8 (visit 2) | 1.647 (0.689) | 1.351 (0.258)

ADVERSE EVENTS:
Groups:
- All Study Particpants: Oral nebivolol 5 mg once daily or Placebo (sugar pill) once dailly. Arms/Groups are combined in this module because the only access to data is a publication that was published before Principal Invesitgator passed away. According to the publication; two participants dropped out because of flu-like symptoms, 2 were lost to follow-up, and 1 dropped out of the study after the initial visit but never took the medication. It is unknown what arm they were in.
Arm/Group | All Study Particpants
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Particpants (N=50)
Flue like symptoms (Infections and infestations) | 1 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes